CLINICAL TRIAL: NCT02213068
Title: Randomized Conversion Of Epstein-Barr Virus (EBV)+ Kidney Transplant Recipients Of Living Or Standard Criteria Donors At Three Months Post Transplantation To Belatacept With MPA Or Belatacept With Low-Dose Tacrolimus (50% Of Dose) Compared To Patients Remaining On Center Specific Standard Therapy Of Tacrolimus And MPA
Brief Title: Belatacept 3 Month Post Transplant Conversion Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lorenzo Gallon (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Lorenzo Gallon, Associate Professor, Northwestern University, Feinberg School of Medicine, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00085274
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2021-09-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Transplant; Failure, Kidney; EBV
Keywords: Kidney; Renal; Transplant; EBV; Immunosuppressants; Belatacept
MeSH Terms: interventions — Abatacept; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- belatacept + MPA (Experimental): subjects continue MPA per SOC, receive bimonthly infusions of belatacept while gradually reducing and then discontinuing tacrolimus:
  Belatacept: 5 mg/kg IV on Day 1, 15, 29, 43, and 57 post-conversion, then monthly thereafter.
  Tacrolimus tapered over one month as follows:
  Days 1- 14: SOC administration Day 15 (~ 2 weeks into study): 40-60% of the previous dose Day 21 (~ 3 weeks into study): 20-30% of the previous dose Day 30 (about 1 month): discontinue
  MPA: administered according to SOC
  Interventions: Drug: belatacept; Drug: MPA
- belatacept + Low-Dose Tac (Active Comparator): Belatacept: 5 mg/kg IV on Day 1, 15, 29, 43, and 57 post-conversion, then monthly thereafter.
  Tacrolimus tapered over one month as follows:
  Days 1- 14: SOC administration Day 15 (~ 2 weeks into study): 10% of the previous dose Day 21 (~ 3 weeks into study): 20% of the previous dose Day 30 (~ 1 month into study): 20% of the previous dose Target trough level ≤ 5 mg per ml of tacrolimus thereafter.
  Interventions: Drug: belatacept; Drug: Tacrolimus
- Tacrolimus + MPA standard treatment regimen (Other): Standard of Care treatment regimen:
  Tacrolimus: administered orally twice daily (BID) The total initial dose of Tacrolimus is given at 0.1 mg/kg in two divided doses to achieve a stable 12-hour trough level of 8 - 12 ng/mL on Days 1 through 30, with dose reduction to achieve a 12-hour trough target of 5 - 10 ng/mL thereafter.
  MPA: dosed orally per package insert beginning on the day of transplantation. Methylprednisolone as sodium succinate is administered as 500 mg IV, 250 mg IV, 125 mg IV, on Days 0, 1, and 2 without corticosteroid taper.
  MPA dose adjustments for gastrointestinal side effects or leukopenia will be made at the discretion of the investigator.
  Interventions: Drug: Tacrolimus; Drug: MPA

INTERVENTIONS:
Drug: belatacept — Please reference Arm description for belatacept + MPA and Arm description for Arm belatacept + Low-Dose Tac for details on this intervention
  Other Names: Belatacept (Nulojix®)
  Arms: belatacept + Low-Dose Tac; belatacept + MPA
Drug: Tacrolimus — Please see Arm Descriptions for both Standard of Care Arm Tacrolimus + MPA standard treatment regimen and belatacept + Low-Dose Tac for details on this intervention
  Other Names: Tacrolimus (Prograf®)
  Arms: Tacrolimus + MPA standard treatment regimen; belatacept + Low-Dose Tac
Drug: MPA — Please see Arm Descriptions for both Standard of Care Arm Tacrolimus + MPA standard treatment regimen and belatacept + MPA for details on this intervention
  Other Names: Mycophenolic Acid (MPA) (Myfortic®)
  Arms: Tacrolimus + MPA standard treatment regimen; belatacept + MPA

SUMMARY:
This study is being done to investigate the impact of changing immunosuppressive medications from tacrolimus (Prograf®) to belatacept (Nulojix®) between three (3) and six (6) months after kidney transplantation. The immune system is the body's defense against infection and other disease. After transplantation, the body sees the new organ as "foreign" and tries to destroy or "reject" it. Immunosuppressive medications help to prevent the immune system from attacking the transplanted organ. The primary purpose of this research study is to evaluate the effects of three (3) different immunosuppressive treatments on rejection in post-transplant kidney recipients. This study will test whether switching from tacrolimus to belatacept will improve long-term kidney function.

Three of the immunosuppressants used in this study- mycophenolic acid (MPA), mycophenolate mofetil (MMF) and tacrolimus- are medications approved by the United States Food and Drug Administration (FDA) to be used after transplant. All of these medications have been routinely used in kidney recipients here at Northwestern University.

Belatacept (the "study drug") has been approved by the FDA for use at the time of transplant. However, the use of belatacept in this study is considered investigational as it has not been FDA approved for use beginning at 3 months after transplant.

This study will involve 51 adult kidney transplant recipients at Northwestern.

DETAILED DESCRIPTION:
Immunosuppressive therapy with the calcineurin inhibitors (CNI) cyclosporine (CsA) and Tacrolimus (Tac), have radically changed the field of organ transplantation. Ironically, although extensively and effectively used for kidney transplantation and other solid organ transplants, CsA and Tac cause important adverse renal side effects: acute and chronic renal dysfunction, hemolytic-uremic syndrome, hypertension, electrolyte disturbances and tubular acidosis. Chronic nephrotoxicity from CNI has been implicated as a principal cause of post-transplant renal dysfunction and it is characterized by an irreversible and progressive tubular atrophy, interstitial fibrosis, and focal hyalinosis of small renal arteries and arterioles. Attempts to minimize CNIs and their known toxicities have been marginally successful due to unacceptable rates of acute rejection and drug toxicity. Patients are converted to alternative immunosuppressive therapy related to CNI side effects including neurotoxicity, nephrotoxicity, cardiovascular (HTN, hyperlipidemia), metabolic (NODAT), and cosmetic side effects. Furthermore, this class of medications is associated also, by blocking Interleukin 2 (IL2) production, with negative impact on regulatory T cells (Tregs) generation (an important subpopulation of T helper cells that has been associated with positive immunomodulation and donor specific hypo-responsiveness).

Until the approval of Belatacept for adult EBV+ renal transplant recipients, there have been limited alternative immunosuppressive agents available to mitigate drug induced renal impairment. The phase III drug trials of Belatacept in combination with MMF and corticosteroids have resulted in significant and sustained improvement in glomerular filtration rate (GFR) at one year through three years post transplant. The overall safety of belatacept compared to cyclosporine in de novo transplant recipients was similar. However, there was an increased rate and severity of early acute rejection and post-transplant lymphoproliferative disorder (PTLD) of the central nervous system in patients treated with belatacept.

In a phase II switch study conducted by Bristol Myers Squibb (BMS), the incidence of acute rejection at 24 months post conversion was similar in patients remaining on CNI (4%) compared to those converted to belatacept (7%). There were no reported cases of post-transplant lymphoproliferative disorder (PTLD) in this patient population as of two years post randomization. However, one belatacept patient from Mexico developed tuberculosis and there were more non-serious fungal infections in the belatacept treated patients.

Mechanistically, CD28 (Cluster of Differentiation 28) and CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) are important for the function of regulatory T cells (Tregs). Belatacept binds to CD80/CD86 (Cluster of Differentiation 80/Cluster of Differentiation 86) ligands on antigen presenting cells (APCs) preventing CD28 to bind with these ligands and deliver the costimulatory signal to activate the T Cell. CTLA-4 is a related receptor expressed on activated T cells that also recognizes CD80/CD86 (Cluster of Differentiation 80/Cluster of Differentiation 86) and is thus termed co-inhibitory. It transmits both cell intrinsic and cell extrinsic negative signals that impair activation.

Investigation of the effect of early conversion to Belatacept at month 3 post-transplant on the subpopulations of T cells and B cells and peripheral blood and allograft biopsy-derived gene expression subpopulation profiles are planned. Optimization of the Belatacept immunosuppressive regimen to achieve good long term renal function and improved graft survival requires understanding the relationships of these cell populations to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria

1. Adult ≥ 18 years of age
2. Male or Female
3. EBV seropositive
4. Recipient of renal transplant from living or deceased donor

Exclusion Criteria

1. Recipients with EBV serostatus negative or unknown
2. History of acute rejection (AR) within 3 months prior to randomization
3. History of positive donor specific antibodies (DSA)
4. History of antibody mediated rejection
5. Positive T-cell lymphocytotoxic cross match
6. Proteinuria >1 g/day or > 0.5 g/day if diabetic
7. Rejection on 3 month post-transplant screening biopsy
8. BK nephropathy at 3 months post-transplant screening biopsy
9. Positive pregnancy test at the time of randomization in female of child bearing potential
10. History of previous transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, The Comprehensive Transplant Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Belatacept + MPA: subjects continue MPA per SOC, receive bimonthly infusions of belatacept while gradually reducing and then discontinuing tacrolimus:
  Belatacept: 5 mg/kg IV on Day 1, 15, 29, 43, and 57 post-conversion, then monthly thereafter.
  Tacrolimus tapered over one month as follows:
  Days 1- 14: SOC administration Day 15 (~ 2 weeks into study): 40-60% of the previous dose Day 21 (~ 3 weeks into study): 20-30% of the previous dose Day 30 (about 1 month): discontinue
  MPA: administered according to SOC
  belatacept: Please reference Arm description for belatacept + MPA and Arm description for Arm belatacept + Low-Dose Tac for details on this intervention
  MPA: Please see Arm Descriptions for both Standard of Care Arm Tacrolimus + MPA standard treatment regimen and belatacept + MPA for details on this intervention
- Belatacept + Low-Dose Tac: Belatacept: 5 mg/kg IV on Day 1, 15, 29, 43, and 57 post-conversion, then monthly thereafter.
  Tacrolimus tapered over one month as follows:
  Days 1- 14: SOC administration Day 15 (~ 2 weeks into study): 10% of the previous dose Day 21 (~ 3 weeks into study): 20% of the previous dose Day 30 (~ 1 month into study): 20% of the previous dose Target trough level ≤ 5 mg per ml of tacrolimus thereafter.
  belatacept: Please reference Arm description for belatacept + MPA and Arm description for Arm belatacept + Low-Dose Tac for details on this intervention
  Tacrolimus: Please see Arm Descriptions for both Standard of Care Arm Tacrolimus + MPA standard treatment regimen and belatacept + Low-Dose Tac for details on this intervention
- Tacrolimus + MPA Standard Treatment Regimen: Standard of Care treatment regimen:
  Tacrolimus: administered orally twice daily (BID) The total initial dose of Tacrolimus is given at 0.1 mg/kg in two divided doses to achieve a stable 12-hour trough level of 8 - 12 ng/mL on Days 1 through 30, with dose reduction to achieve a 12-hour trough target of 5 - 10 ng/mL thereafter.
  MPA: dosed orally per package insert beginning on the day of transplantation. Methylprednisolone as sodium succinate is administered as 500 mg IV, 250 mg IV, 125 mg IV, on Days 0, 1, and 2 without corticosteroid taper.
  MPA dose adjustments for gastrointestinal side effects or leukopenia will be made at the discretion of the investigator.
  Tacrolimus: Please see Arm Descriptions for both Standard of Care Arm Tacrolimus + MPA standard treatment regimen and belatacept + Low-Dose Tac for details on this intervention
  MPA: Please see Arm Descriptions for both Standard of Care Arm Tacrolimus + MPA standard treatment regimen and belatacept + MPA for details on this intervention
Period: Overall Study
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen
Started | 9 | 8 | 10
Completed | 9 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen | Total
Number analyzed (Participants) | 9 | 8 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (16.21) | 49.75 (13.33) | 49.70 (13.53) | 48.81 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 11
  Male | 7 | 3 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 5 | 9
  Not Hispanic or Latino | 1 | 1 | 1 | 3
  Unknown or Not Reported | 5 | 6 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 4 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 10 | 27
Incidence of Delayed Graft Function [Count of Participants; unit: Participants] — Delayed graft function is defined as the need for hemodialysis during the first week post-transplant.
  Participants | 0 | 0 | 1 | 1
Incidence of Diabetes [Count of Participants; unit: Participants] | 0 | 2 | 3 | 5
Incidence of Hypertension [Count of Participants; unit: Participants] | 8 | 6 | 10 | 24
Positive Cross-Match [Count of Participants; unit: Participants] — T and B cell crossmatch is used pre-transplant to measure pre-sensitizing events against the kidney transplant. In other words, a positive cross-match prior to transplantation may indicate worse outcomes for the kidney graft survival.
  Participants | 0 | 0 | 0 | 0
Baseline Kidney Function as eGFR [Mean (Standard Deviation); unit: mL/min/1.73m2] — eGFR = estimated glomerular filtration rate.
  mL/min/1.73m2 | 67.33 (17.89) | 67.75 (20.01) | 70.70 (20.70) | 70.19 (20.19)

OUTCOME MEASURES:

1. Primary Outcome: Change in eGFR (MDRD) at 2 Years Post-transplant Compared to Baseline at Month 3 (Conversion)
Description: To assess change in renal function by calculated (MDRD) GFR of adult EBV seropositive renal transplant recipients of living or standard criteria donors converted from Tacrolimus to Belatacept or low dose Tacrolimus with Belatacept at three months post-operatively compared to renal transplant recipients randomized to remain on standard dose Tacrolimus and MPA for maintenance therapy at 2 years post-transplantation
Time Frame: 2 years
Measure: Mean (Standard Error); unit: mL/min/1.73m2
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen
Number analyzed (Participants) | 9 | 8 | 10
mL/min/1.73m2 | -5.44 (5.43) | 8.08 (5.74) | -0.38 (3.94)

2. Primary Outcome: Acute Rejection
Description: Number of Participants with Acute Rejection (AR). AR is defined as allograft dysfunctions in the setting of recipient immune system engaging an allo-response against the kidney transplant.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen
Number analyzed (Participants) | 9 | 8 | 10
Participants | 4 | 0 | 2

3. Primary Outcome: Graft Survival
Description: Number of Subjects with a functioning Graft
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen
Number analyzed (Participants) | 9 | 8 | 10
Participants | 8 | 8 | 10

4. Primary Outcome: Patient Survival
Description: Number of Subjects alive at the end of 24 months
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen
Number analyzed (Participants) | 9 | 8 | 10
Participants | 9 | 7 | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Belatacept + MPA | Belatacept + Low-Dose Tac | Tacrolimus + MPA Standard Treatment Regimen
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/8 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/8 | 1/10
Other Adverse Events (participants affected / at risk) | 6/9 | 7/8 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept + MPA (N=9) | Belatacept + Low-Dose Tac (N=8) | Tacrolimus + MPA Standard Treatment Regimen (N=10)
Death (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Patient developed pneumonia with overwhelming sepsis. Not thought to be related to study intervention.
Death (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) — Diabetic ketoacidosis
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — SCC skin cancer removed from nose
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept + MPA (N=9) | Belatacept + Low-Dose Tac (N=8) | Tacrolimus + MPA Standard Treatment Regimen (N=10)
CMV (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
BK infections (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT02213068/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT02213068/ICF_001.pdf